CLINICAL TRIAL: NCT00258011
Title: A Safety Confirmatory Study of JC0498 (Laronidase) in Mucopolysaccharidosis I (MPS I) Patients
Brief Title: Study of Aldurazyme® Replacement Therapy in Patients With Mucopolysaccharidosis I (MPS I) Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: BioMarin/Genzyme LLC (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALID02205
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Results first posted 2009-02-12 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: Mucopolysaccharidosis I; Hurler Syndrome; Hurler-Scheie Syndrome; Scheie Syndrome
Keywords: MPS I Disease
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — Iduronidase

ARMS (1):
- Aldurazyme (laronidase) treatment (Experimental): Patients received weekly infusions of JC0498 (laronidase) at an intravenous dose of 100 Units/kg (0.58 mg/kg) body weight for up to 73 weeks.
  Interventions: Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase)

INTERVENTIONS:
Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase) — 0.58 mg/kg every week

SUMMARY:
This is a multi-center, open label, study conducted to evaluate the safety of laronidase administered by intravenous drip infusion in Japanese patients with MPS I disease.

Following baseline evaluation, patients will receive weekly infusions of JC0498 at an intravenous dose of 100 units/kg. Patient safety will be monitored continuously throughout the trial. In addition, the effects of JC0498 treatment in this patient population will be assessed by periodically evaluating aspects of MPS I disease in patients at scheduled intervals over the duration of the trial.

Since patients may be eligible for the trial if they have received JC0498, a portion of the data may be captured retrospectively and recorded onto the case report forms (CRFs).

This study represents the first good clinical practice (GCP) effort to characterize MPS I in the Japanese population and evaluate the effects of JC0498 on disease manifestations.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent of the patient or written informed consent of the parent(s) or the legal guardian(s), depending on the age of the patient, is required prior to any protocol-related procedures being performed; this includes information regarding hematopoietic stem cell transplantation (HSCT) in order to assure that the guardian(s) is fully informed regarding the risks and benefits of this alternative treatment for patients eligible for the trial and who have severe manifestations of MPS I with neurodegeneration.
* Have a clinical diagnosis of MPS, confirmed by measurable clinical signs and symptoms of MPS I.
* Have confirmed iduronidase deficiency with a leukocyte alpha-L-iduronidase enzyme activity level of less than 10.0% of the lower limit of the normal range of the measuring laboratory (SRL)

Exclusion Criteria:

* The patient is under consideration for or has previously undergone hematopoietic stem cell transplantation.
* The patient has acute hydrocephalus at the time of enrollment.
* The patient has a clinically significant organic disease (with the exception of symptoms relating to MPS I) including: cardiovascular, hepatic, pulmonary, neurologic, or renal disease, other serious intercurrent illness, or extenuating circumstances that, in the opinion of the Investigator, would preclude participation in the trial or potentially decrease survival.
* The patient has received any investigational product within 30 days prior to trial enrollment (exception: JC0498).
* The patient has known severe hypersensitivity to JC0498 or components of the delivery solution.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-12; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigetoyo Oguri, Study Director — Corp. GCP Compliance - Clinical Affairs, Genzyme Japan K.K.
Locations (2):
- Japan (2):
  - Osaka City University Hospital, Osaka
  - National Center for Child Health and Development, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Aldurazyme (Laronidase) Treatment: Patients received weekly infusions of Aldurazyme (laronidase) at an intravenous dose of 100 Units/kg (0.58 mg/kg) body weight (labeled dose) for up to 73 weeks.
Period: Overall Study
Arm/Group | Aldurazyme (Laronidase) Treatment
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aldurazyme (Laronidase) Treatment
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian (Japanese) | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety Evaluation
Description: Overall Safety Summary of Adverse Events (AEs) during Treatment Safety assessment was based on the incidence of AE reports.
Time Frame: Up to 73 Weeks
Population: The study enrolled eligible MPS I patients prior to marketing authorization in Japan. The analysis was intention to treat.
Measure: Number; unit: participants
Arm/Group | Aldurazyme (Laronidase) Treatment
Number analyzed (Participants) | 3
participants
  Having Adverse Events (AEs) | 3 [-81.1 to -60.6]
  Having drug related AEs | 0
  Discontinuations due to AEs | 0
  Having Serious AEs | 1
  Having Severe AEs | 1
  Deaths | 0
  Having infusion-associated reactions | 0

2. Secondary Outcome: Urinary Glycosaminoglycan (GAG) Excretion
Description: Percentage change in the concentration of GAG relative to creatinine in urine (ug GAG/mg creatinine) from baseline to last study visit. Greater decrease indicates greater response.
Time Frame: Up to 73 Weeks
Population: The study enrolled eligible MPS I patients prior to marketing authorization in Japan. The analysis was intention to treat.>
  * 1 patient final visit = Week 73; 1 patient final visit = Week 32; 1 patient final visit = Week 10
Measure: Mean (Standard Deviation); unit: percent change in concentration of GAG
Arm/Group | Aldurazyme (Laronidase) Treatment
Number analyzed (Participants) | 3
percent change in concentration of GAG
  Baseline (3 patients analyzed) | 0 (0)
  Week 4 (3 patients analyzed) | -68.0 (12.76)
  Week 8 (3 patients analyzed) | -69.9 (7.98)
  Week 12 (2 patients analyzed) | -74.6 (11.47)
  Week 16 (2 patients analyzed) | -71.0 (9.40)
  Week 20 (2 patients analyzed) | -60.6 (12.85)
  Week 26 (2 patients analyzed) | -71.5 (5.84)
  Week 30 (2 patients analyzed) | -75.2 (10.65)
  Week 34 (1 patients analyzed) | -77.7 (0)
  Week 38 (1 patients analyzed) | -69.9 (0)
  Week 42 (1 patients analyzed) | -78.0 (0)
  Week 46 (1 patients analyzed) | -67.9 (0)
  Week 52 (1 patients analyzed) | -77.0 (0)
  Week 64 (1 patients analyzed) | -81.1 (0)
  Final Examination * (3 patients analyzed) | -69.7 (20.23)

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Groups:
- Aldurazyme: Aldurazyme
Arm/Group | Aldurazyme
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aldurazyme (N=3)
Bronchitis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aldurazyme (N=3)
Conjunctivitis (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Catheter related complication (General disorders) | 1
Catheter site erythema (General disorders) | 1
Catheter site pruritus (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Otitis media (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Oxygen saturation decreased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 1
Insomnia (Psychiatric disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Heat rash (Skin and subcutaneous tissue disorders) | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Pallor (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the rarity of the disease, this study is limited by its small sample size, lack of a control group and patients had variable treatment durations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.